CLINICAL TRIAL: NCT01949467
Title: Prospective, Comparative (5 Groups), Non-randomized, Multicenter, Physiopathological Study, Evaluating Pharmacokinetic Characteristics of Serum Hepcidin Level in Response to Iron Oral Intake in Order to Evaluate Their Interest to Discriminate Patients With Dysmetabolic Hepatosiderosis or Ferroportin Disease.
Brief Title: Analysis of the Modulation of Serum Hepcidin Level in Response to Iron Oral Intake: Potential Interest for the Differential Diagnosis Between Ferroportin Disease and Dysmetabolic Hepatosiderosis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FERHEP
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2018-08

CONDITIONS: Hemochromatosis, Type 4; Ferroportin Disease; Dysmetabolic Hepatosiderosis; Diagnosis
Keywords: ferroportin disease; dysmetabolic hepatosiderosis; genetic hemochromatosis; hyperferritinemia; hepcidin; iron fumarate; physiopathological study; diagnosis; HFE gene; TRF2 gene; iron parameters; divalent cations
MeSH Terms: conditions — Hemochromatosis, type 4; Disease; Hemochromatosis; Hyperferritinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- TDHS (Other): 20 Patients with Treated Dysmetabolic Hepatosiderosis (TDHS)
  Interventions: Drug: iron fumarate
- UDHS (Other): 20 patients with untreated Dysmetabolic Hepatosiderosis (UDHS)
  Interventions: Drug: iron fumarate
- TFPD (Other): 20 patients with treated Ferroportin Disease (TFPD)
  Interventions: Drug: iron fumarate
- UFPD (Other): 20 patients with untreated Ferroportin Disease (UFPD)
  Interventions: Drug: iron fumarate
- HV (Other): 20 Healthy volunteers (HV) patients
  Interventions: Drug: iron fumarate

INTERVENTIONS:
Drug: iron fumarate — All patients will receive a tablet of 66mg of iron, in the form of iron fumarate (Fumafer®) with 50 ml water.

SUMMARY:
The diagnosis of iron overload is a common problem. It is important to optimize the diagnosis to ensure support for patients and their relatives especially regarding genetic disease.

Iron overload revealed by a high level of serum ferritin and confirmed by the presence of an excessive amount of iron in the liver is a frequent situation. In a lot of case there is no increase in serum iron and transferrin saturation. This situation may arise in particular in patients with:

* a genetic iron overload related to mutation in the ferroportine gene, leading to a ferroportin disease. The diagnosis is based on the sequencing of the gene,
* a dysmetabolic hepatosiderosis, the most frequent situation , where iron overload is associated with abnormalities in the metabolism of carbohydrates and fats, whereas no genetic cause is identified.

However, patients often have similar biological signs and despite the implementation of strict algorithm regarding the diagnostic procedure, it appears that a large number of patients are tested for the mutation in the ferroportin gene, and that mutation is not found in most cases. It is therefore essential to optimize the diagnosis process by introducing additional criteria.

The investigators' hypothesis, based on the known elements, is that the response to a single dose of iron will modulate differently the iron parameters measured in serum, including hepcidin level which controls iron metabolism and metals associated with iron. This could be helpful for diagnosis procedure in patients with ferroportin disease or dysmetabolic hepatosiderosis.

DETAILED DESCRIPTION:
The quantification of serum hepcidin level is a potential method of investigation in iron metabolism disorders. However, apart from some extreme situations, the assay achieved solely is not helpful. This is due to the varying levels encountered from one subject to another for the same disease. This is related to the facts that values considered to be normal cover a wide range and that a value obtained for a given patient at a given time, can be influenced by many factors.

It has been reported that a a single oral iron dose induced an increase of serum hepcidin level in healthy subjects which is abolished in subjects with genetic hemochromatosis linked to insufficient hepcidin expression related to mutations in the HFE or TFR2 genes.

In patients with a dysmetabolic hepatosiderosis, it was suggested that the expected hepcidinemia increase found after an iron intake was altered, likely due to a slight inflammatory signal responsible for hepcidin induction.

The investigators hypothesize that a dynamic response of iron parameters, including modulation of hepcidin level, to an iron intake will allow to discriminate patients with ferroportin disease or dysmetabolic hepatosiderosis, situations whose clinicobiological presentation is often confusing.

Thus, the three objectives in this study will be :

1. To define pharmacokinetic characteristics of serum hepcidin in response to iron oral intake and to determine the ability of this pharmacokinetic to discriminate dysmetabolic hepatosiderosis and ferroportin disease.
2. To correlate amplitude of this response to the iron parameters modulation
3. To correlate amplitude of this response to the concentration of divalent cations whose metabolism uses common genes to those involved in iron metabolism.

ELIGIBILITY:
Inclusion Criteria for patients:

* Man or woman older than 18 years
* Subject having a liver iron overload greater than or equal to 100 umol /g dry liver weight, confirmed by MRI (done performed with body antenna and complete deactivation of the surface antenna) and / or by biochemical assay on liver biopsy, and related to dysmetabolic hepatosiderosis or ferroportin disease.

  * The ferroportin disease will be retained when patients will present an hyperferritinemia without elevated transferrin saturation and a heterozygote mutation in the gene encoding ferroportin.
  * A dysmetabolic hepatosiderosis will be retained following the usual diagnostic investigation including sequencing of the gene for ferroportin (mutation proven negative), if patients do not show any other cause of iron overload and hyperferritinemia is not related to excessive alcohol intake, non-metabolic liver cytolysis (hepatitis C virus, wilson, autoimmune hepatitis, ...), hemolysis, or inflammatory syndrome.
* Status towards the iron-depletive treatment : either no venesection performed (Dysmetabolic HepatoSiderosis and Ferroportin disease groups) or attack iron depletive treatment completed (Treated Dysmetabolic Hepatosiderosis and Treated Ferroportin Disease groups) with ferritin level less than 100 ng / ml, without anemia and with no venesection in the two last months.
* Having given a free and informed consent in writing
* Affiliate to the social security system.

Exclusion Criteria for patients:

* Alcohol consumption greater than 30g/d
* Chronic inflammatory disease.
* HIV, HCV or HBV Infection.
* Blood donation in the last three months.
* Infection during the previous seven days before testing
* Staying in altitude (>1500 m) dating less than 2 months
* Night occupation or shift work.
* Pregnancy
* Exclusion period in the national register of persons suitable for biomedical research.
* Protected adults (judicial protection, guardianship and trusteeship) and persons deprived of liberty

Inclusion criteria for healthy volunteers:

* Man or woman older than 18 years.
* Body Mass Index between 18 and 25 kg/m².
* Non smoker or quit smoking for more than 6 months
* Examen clinique normal. Normal clinical examination
* Normal ECG.
* Normal values for routine laboratory tests : serum iron, tranferrin saturation, CBC, ferritin, blood cell count C-reactive protein, AST, ALT, GGT, HDL and LDL cholesterol, triglycerides.
* Having given a free and informed consent in writing
* Affiliate or beneficiary to the social security system.

Exclusion criteria for healthy volunteers :

* Progressive and/or chronic disease.
* Infection during the previous seven days before testing
* Drug use under 6 months.
* Alcohol consumption greater than 30g/d
* Medication ongoing or stopped from less than a week (except contraceptives).
* History of blood transfusion or martial treatment.
* Staying in altitude (>1500 m) dating less than 2 months
* Night occupation or shift work.
* Known infection by hepatitis B or C.
* Positive serology for HIV.
* Blood donation in the last three months.
* Pregnancy.
* Exclusion period in the national register of persons suitable for biomedical research.
* Protected adults (judicial protection, guardianship and trusteeship) and persons deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
hepcidemia rate | Day 1
  The primary endpoint is the maximum variation, of hepcidemia rate (Δmax) after iron oral intake. This variation will be compared between the different groups of included subjects

SECONDARY OUTCOMES:
ratios between serum hepcidin level and iron parameters | Day 1
  Differential modulation, induced by the iron intake, of ratios between serum hepcidin level and iron parameters (serum iron, transferrin, ferritin) between the different groups.
serum level of other divalent cations | day 1
  Modulation of serum level of other divalent cations.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Limoges, Limoges
  - CHU Montpellier, Montpellier
  - CHU Pontchaillou, Rennes